CLINICAL TRIAL: NCT03187795
Title: Efficacy and Tolerability of Mirabegron Compared to Oxybutynin Chloride Immediate Release for Neurogenic Detrusor Overactivity in Persons With Chronic Spinal Cord Injury: A Randomized, Double-Blind, Controlled, Cross-Over Clinical Trial
Brief Title: Mirabegron and Oxybutynin Safety and Efficacy Trial in Spinal Cord Injury
Acronym: MOSET-SCI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Trevor Dyson-Hudson, M.D., Director, Spinal Cord Injury Research, Kessler Foundation
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D-961-17
Record Dates: First submitted 2017-06-12; First posted 2017-06-15 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Spinal Cord Injuries; Urinary Bladder, Neurogenic
Keywords: Spinal Cord Injuries; Randomized Controlled Trial; Neurogenic Bladder; Rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Bladder, Neurogenic | interventions — oxybutynin; mirabegron

STUDY DESIGN:
Intervention Model Description: After a two-day washout period, participants will be randomly assigned to one of two treatment groups: 1) an escalating dose of mirabegron for 6 weeks (25 mg once daily plus two placebo pills for 2 weeks, followed by 50 mg once daily plus 2 placebo pills for 4 weeks); or 2) Oxybutynin IR (5 mg orally three times daily) for 6 weeks. All participants will then be switched to the opposite study treatment for 6 weeks. Assessments will be performed at Baseline, Week 6 (completion of first study medication and prior to administration of second study medication), and Week 12 (completion of second study medication).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study investigators, participants, and assessors will be blind to group assignment. Blinding code will only be broken in emergency situations for reasons of subject safety, where knowledge of the treatment administered is necessary for the treatment of the adverse event under Good Clinical Practices (GCPs), or when required by local regulatory authorities.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Oxybutynin chloride IR then Mirabegron (Experimental): Subjects randomized to this group will receive oxybutynin IR (5 mg three times daily) for 6 weeks. After the initial 6 weeks, subjects in this group will then be switched to an escalating dose of mirabegron for 6 weeks (25 mg once daily for 2 weeks, followed by 50 mg once daily for 4 weeks; Note: two placebo daily will be included with mirabegron once daily to match the frequency of dosing to oxybutynin IR three times daily).
  Interventions: Drug: Oxybutynin Chloride IR; Drug: Mirabegron
- Mirabegron then Oxybutynin chloride IR (Experimental): Subjects randomized to this group will receive an escalating dose of mirabegron for 6 weeks (25 mg once daily for 2 weeks, followed by 50 mg once daily for 4 weeks; Note: two placebo daily will be included with mirabegron once daily to match the frequency of dosing to oxybutynin IR three times daily). After the initial 6 weeks, subjects in this group will then be switched to receive oxybutynin IR (5 mg three times daily) for 6 weeks
  Interventions: Drug: Oxybutynin Chloride IR; Drug: Mirabegron

INTERVENTIONS:
Drug: Oxybutynin Chloride IR — Oxybutynin chloride immediate release (IR) 5 mg three times daily for 6 weeks
  Other Names: Ditropan
Drug: Mirabegron — Mirabegron 25 mg tablet once daily for 2 weeks, followed by mirabegron 50 mg once daily for 4 weeks (Note: Placebo twice daily will be included with mirabegron once daily to match the three-time daily dosing of oxybutynin IR in the other intervention).
  Other Names: Myrbetriq

SUMMARY:
The purpose of this research study is to determine the effectiveness and safety of mirabegron compared to oxybutynin chloride immediate release (oxybutynin IR) for a condition called neurogenic detrusor overactivity in individuals with chronic spinal cord injury (SCI).

DETAILED DESCRIPTION:
Neurogenic detrusor overactivity or "NDO" is common in people with spinal cord injury (SCI) and is a medical condition characterized by involuntary urinary bladder contractions. These bladder contractions can cause episodes of urinary incontinence (involuntary urine leakage) and/or high bladder pressures that can lead to poor drainage from the kidneys and urinary tract infections (UTIs).

Neurogenic detrusor overactivity is most commonly treated with a medication called oxybutynin (Ditropan); however, this medication is associated with side effects such as dry mouth and constipation. Mirabegron (Myrbetriq) is a newer medication approved by the Food and Drug Administration for the treatment of overactive bladder that does not cause dry mouth or constipation; however, its use in persons with SCI is investigational.

The purpose of this research study is to determine the effectiveness and safety of mirabegron compared to oxybutynin chloride immediate release (oxybutynin IR) for neurogenic detrusor overactivity in individuals with SCI.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a neurological impairment secondary to a traumatic spinal cord injury that occurred at least twelve (12) months prior to the screening visit.
* The injury is classified as complete or incomplete (AIS grade A-D) and the neurological level of the injury is above T12.
* The subject's method of bladder management is intermittent catheterization (IC) or indwelling catheter (transurethral or suprapubic).
* There is urodynamic documentation of neurogenic detrusor overactivity (NDO).
* The subject is on a stable dose of oxybutynin IR three times daily.
* The subject is able and willing to comply with the study protocol, including availability for all scheduled clinic visits and locomotor training sessions.
* The subject is able to and has voluntarily given informed consent prior to the performance of any study-specific procedures.

Exclusion Criteria:

* The subject has taken mirabegron within one month of the Screening Visit.
* The subject has received a botulinum toxin injection to the bladder within one year of the Screening Visit.
* The subject is allergic to mirabegron.
* The subject has a history of uncontrolled autonomic dysreflexia or significant autonomic dysreflexia on urodynamics (systolic BP≥150 mm/Hg).
* The subject has a known history of significant anatomical problems of the upper tracts, including hydronephrosis, kidney stones, or ureteropelvic junction obstruction.
* The subject has a known history or treatment for a non-neurogenic bladder or prostate problem (prostate cancer, bladder cancer).
* The subject has recurrent UTIs, defined as a UTI more than every three months.
* The subject has untreated Grade 3 or above vesicoureteral reflux.
* If female, the subject is pregnant (documented by a urine pregnancy test) or breastfeeding.
* The subject has taken another investigational drug within 30 days before screening.
* The subject has a medical condition that might pose a safety issue or would interfere with interpretation of study results or study conduct.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2019-04-03 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in cystometric bladder capacity during filing cystometry | Week 6 and Week 12
  The cystometric bladder capacity is the bladder volume (ml) at the end of the filling cystometrogram, when 'permission to void' is usually given.

SECONDARY OUTCOMES:
Change in detrusor leak point pressure | Week 6 and Week 12
  The detrusor leak point pressure (cm H2O) is defined as the lowest detrusor pressure at which urine leakage occurs in the absence of either a detrusor contraction or increased abdominal pressure.
Change in maximum detrusor pressure | Week 6 and Week 12
  Maximum detrusor pressure (ml/cm H2O) as the name implies, is the maximum detrusor pressure during filling cystometry.
Change in bladder compliance during filling cystometry | Week 6 and Week 12
  Bladder compliance during filling cystometry (ml/cm H2O) is the relationship between change in bladder volume and change in detrusor pressure and is calculated by dividing the volume change (ΔV) by the change in detrusor pressure (Δρdet) during that change in bladder volume (C= ΔV/Δρdet).
Change in post-void residual volume | Week 6 and Week 12
  The post-void residual volume (ml) is defined as the volume of urine left in the bladder at the end of micturition1 and is recommended as a core urodynamic outcome measure in SCI.
Change on International Lower Urinary Tract Function Basic Spinal Cord Injury (SCI) Data Set | Week 6 and Week 12
  The purpose of the Lower Urinary Tract Function Basic Data Set for Spinal Cord Injury (SCI) individuals is to standardize the collection and reporting of information on the lower urinary tract and to make it possible to evaluate and compare results from various published studies.
Change on Bowel Function Measures - International SCI Bowel Function Basic & Extended Data Sets | Week 6 and Week 12
  The International Bowel Function Basic and Extended SCI Data Sets present a standardized format for the collection and reporting of an extended amount of information on bowel function in persons with SCI.
Change in California Verbal Learning Test - II (CVLT) scores | Week 6 and Week 12
  Memory will be assessed by the California Verbal Learning Test - II (CVLT). It consists of a list of 16 words from 4 semantic categories presented orally over 5 trials and includes a 20 minute delayed recall trial as well as a recognition trial.
Change in Symbol Digit Modalities Test oral version (SDMT) scores | Week 6 and Week 12
  Processing speed will be assessed by the Symbol Digit Modalities Test oral version.
Wechsler Test of Adult Reading (WTAR) score | Screening Visit
  The Wechsler Test of Adult Reading will be administered to provide an estimate of verbal intelligence for later use as a covariate in the analyses of the cognitive outcomes. The WTAR is composed of 50 irregularly spelled words and takes approximately 10 minutes to complete.
Change in Qualiveen scores | Week 6 and Week 12
  The Qualiveen was developed as a condition-specific QOL measure for individuals with SCI. It consists of 30 items focusing on four aspects of individuals' lives related to their urinary problems: bother with limitations, frequency of limitations, fears, and feelings.
Change in SCI-QOL Bowel & Bladder Management Difficulties scores | Week 6 and Week 12
  The SCI-QOL Bladder Management Difficulties and SCI-QOL Bowel Management Difficulties were developed as QOL measure for individuals with SCI and are part of the SCI-QOL measurement system.
Change in Subject Global Impression (SGI) of Change score | Week 6 and Week 12
  The SGI of change is a subject-rated instrument that measures change in the subject's overall status on a 7-point scale.
Change in Clinician Global Impression (CGI) of Change score | Week 6 and Week 12
  The study physician will rate on a 7-point scale the subject's overall clinical condition following treatment as compared to that at baseline.

OTHER OUTCOMES:
Adverse Event Case Report Form | Every two weeks for 12 weeks
  Adverse experience(s) will be recorded on the Adverse Event Case Report Form, including the date and time of onset, severity, the relationship to study intervention, the date of resolution, the action taken, and the outcome of the adverse experience. The responsible physician will make a causality assessment for every adverse experience.
Side Effects Record | Every two weeks for 12 weeks
  Participants will be provided a list of side-effects associated with oxybutynin and mirabegron treatment. Three lines marked "other" for open-choice responses will accompany the selection of options for forced-choice side-effects. Participants will rate the severity (visual analog scale (VAS); 0-100) and frequency ("never", "occasionally", "sometimes", "often" or "always") of side effects for each of the forced and open choice answers. Severity and frequency of side-effects will be rated by participants every 2 weeks during the intervention part of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Todd A. Linsenmeyer, M.D., Principal Investigator — Kessler Institute for Rehabilitation; Steven C. Kirshblum, M.D., Principal Investigator — Kessler Institute for Rehabilitation; Trevor A. Dyson-Hudson, M.D., Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Institute for Rehabilitation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided